CLINICAL TRIAL: NCT00002083
Title: Intranasal Peptide T in the Treatment of Painful Peripheral Neuropathy of AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Peptides (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 115A; 01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-03

CONDITIONS: HIV Infections; Peripheral Nervous System Disease
Keywords: Peptide T; HIV-1; Administration, Intranasal; Acquired Immunodeficiency Syndrome; Peripheral Nervous System Diseases
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Acquired Immunodeficiency Syndrome | interventions — Peptide T

INTERVENTIONS:
Drug: Peptide T

SUMMARY:
To compare the effects of intranasal peptide T and placebo in the treatment of painful peripheral neuropathy associated with human immunodeficiency virus (HIV) infection.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV-1 infection.
* CD4 count < 500 cells/mm3.
* HIV-1-associated distal symmetrical polyneuropathy, with peripheral neuropathy present for at least 6 weeks prior to study entry.
* Pain severity of at least 8 on an analog scale.
* Prior zidovudine therapy for at least the previous 3 months (unless patient has shown intolerance to zidovudine).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Neuropathy due to any other cause besides HIV infection.
* Any symptom consistent with a new or active underlying opportunistic infection or malignancy that could interfere with the evaluation of neuropathy.
* Clinical evidence of new or active CNS disease, potentially from opportunistic infection or neoplasm resulting from HIV infections, that could interfere with the evaluation of neuropathy.
* Other CNS disease (e.g., myelopathy) that could complicate the evaluation of neuropathy.
* Active life-threatening illness other than AIDS.

Concurrent Medication:

Excluded:

* Dapsone.
* Hydralazine.
* Isoniazid (INH).
* Current use of tricyclic antidepressants, anticonvulsants, or clonidine unless the patient has used the drug without a change in dose for at least 3 months prior to study entry.
* Narcotics, unless the patient has been using them for at least 6 weeks prior to study entry.

Prior Medication:

Excluded:

* ddI or ddC in the past 8 weeks.
* Prior peptide T.
* Prior tricyclic antidepressants, anticonvulsants, or clonidine unless they have been used for at least 3 months without change in dose.
* Other investigational drugs within the past 30 days.

Required:

* Zidovudine (if intolerance not demonstrated).

Required:

* Zidovudine for at least the previous 3 months (unless patient has demonstrated intolerance to zidovudine).

Chronic alcohol abuse, or current abuse of psychoactive recreational drugs as defined in DSM IIIR. Patients who may be regarded as unreliable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Univ of Miami School of Medicine, Miami, Florida
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Klingenstein Clinical Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York

REFERENCES:
- [Background] MacFadden DK, Doob PR. Role of peptide T in palliation of HIV-1-related painful peripheral neuropathy. Int Conf AIDS. 1991 Jun 16-21;7(2):225 (abstract no WB2173)